CLINICAL TRIAL: NCT05555641
Title: Efficacy and Safety of Nafamostat Mesylate for VV-ECMO Anticoagulation: a Randomized, Single-blind, Multicenter Exploratory, Heparin-controlled Trial
Brief Title: Efficacy and Safety of Nafamostat Mesylate for VV-ECMO Anticoagulation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaobo Yang, MD (Other)
Responsible Party: Sponsor-Investigator, Xiaobo Yang, MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMST20211022
Record Dates: First submitted 2022-09-16; First posted 2022-09-27 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Critical Illness; Anticoagulation
Keywords: Extracorporeal Membrane Oxygenation; Nafamostat mesylate; Unfractionated heparin; Anticoagulation
MeSH Terms: conditions — Critical Illness | interventions — nafamostat; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nafamostat Mesylate (Experimental): VV-ECMO patients were given continuous anticoagulation with nafamostat mesylate, coagulation function was monitored every 6 hours, and APTT was maintained at 1-1.75 times the upper limit of normal detection until reaching the study endpoints, including 14 days after enrollment, 24 hours after withdrawal from ECMO, or any switch to ECMO mode during ECMO treatment.
  Interventions: Drug: Nafamostat Mesylate
- Unfractionated Heparin (Active Comparator): VV-ECMO patients were given continuous anticoagulation with unfractionated heparin, coagulation function was monitored every 6 hours, and APTT was maintained at 1-1.75 times the upper limit of normal detection until reaching the study endpoints, including 14 days after enrollment, 24 hours after withdrawal from ECMO, or any switch to ECMO mode during ECMO treatment.
  Interventions: Drug: Unfractionated Heparin

INTERVENTIONS:
Drug: Nafamostat Mesylate — ECMO patients were given continuous anticoagulation with nafamostat mesylate, coagulation function was monitored every 6 hours, and APTT was maintained at 1-1.75 times the upper limit of normal detection until reaching the study endpoints, including 14 days after enrollment, 24 hours after withdrawal from ECMO, or any switch to ECMO mode during ECMO treatment.
  Arms: Nafamostat Mesylate
Drug: Unfractionated Heparin — ECMO patients were given continuous anticoagulation with unfractionated heparin, coagulation function was monitored every 6 hours, and APTT was maintained at 1-1.75 times the upper limit of normal detection until reaching the study endpoints, including 14 days after enrollment, 24 hours after withdrawal from ECMO, or any switch to ECMO mode during ECMO treatment.
  Arms: Unfractionated Heparin

SUMMARY:
The purpose of this study was to compare the efficacy and safety of nafamostat mesylate and unfractionated heparin during ECMO anticoagulation in critically ill patients.

DETAILED DESCRIPTION:
During ECMO treatment, nafamostat mesylate and unfractionated heparin were randomly administered for continuous anticoagulation, respectively, and the incidence of bleeding and thrombotic complications during anticoagulation was compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >= 18 and <= 80 years;
* Successfully established ECMO (VA/VV) treatment by percutaneous puncture due to cardiogenic shock or respiratory failure;
* Anticoagulation required during ECMO treatment; Before the establishment of ECMO, the APTT test value was within the normal range, and the platelets were not less than 80G/L;
* Within 48 hours of ECMO establishment, APTT test results were between 1 and 1.75 times the upper limit of normal, PLT>80 G/L, and no serious bleeding and thrombosis;
* Sign the informed consent.

Exclusion Criteria:

* Pregnant;
* Bleeding risk or active bleeding;
* Pre-existing diseases requiring long-term anticoagulation before ECMO: pulmonary embolism, deep vein thrombosis, intraventricular thrombosis, atrial fibrillation, etc.;
* Long-term use of anticoagulants before ECMO;
* Antiplatelet drugs were used before ECMO;
* Allergy to heparin, nafamostat mesylate;
* Repeated puncture at the same site for more than 3 times;
* Expected ECMO treatment time < 3 days;
* Patients with an expected survival period of less than 48 hours;
* Patients undergoing extracorporeal cardiopulmonary resuscitation;
* Burn patients; Blood purification treatment using polyacrylonitrile membrane filter;
* Heterozygous ECMO mode or ECMO therapy solely for CO2 removal;
* Other reasons that the investigator considers inappropriate for inclusion;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe bleeding during ECMO | Up to 14 days.
  The ratio of the number of patients with severe bleeding complications to the total number of cases in each group.

SECONDARY OUTCOMES:
Incidence of thrombosis during ECMO | Up to 14 days.
  The ratio of the number of patients with thrombosis complication to the number of cases in each group.
Bleeding-free days during ECMO | Up to 14 days.
  Days without bleeding complications
Oxygenator replacement frequency | Up to 14 days.
  Oxygenator replacement frequency and average number of replacements per patient;
The incidence of ECMO dysfunction | Up to 14 days.
  The ratio of the number of cases with ECMO dysfunction in each group to the total number of cases.
The average amount of red, plasma, cryoprecipitate, fibrinogen, and platelets per person per ECMO day | Up to 14 days.
  Average blood transfusion volume per ECMO day, including red blood cells, plasma, cryoprecipitate, fibrinogen, and platelets.
The compliance rate of APTT test results | Up to 14 days.
  The ratio of the number of APTT tests that met the requirements to the total number of APTT tests during ECMO.
Case fatality rate within 28 days | Up to 28 days.
  After follow-up, the fatality rates of all enrolled patients in each group within 28 days of the study began.
In-hospital mortality | Through study completion, an average of 2 months.
  The fatality rates of all enrolled patients in each group during hospitalization.
Average length of ICU stay. | Through study completion, an average of 2 months.
  Average number of days in ICU for each group of patients.
Average length of hospital stay | Through study completion, an average of 2 months.
  The mean of the total hospitalization days for each group of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided